CLINICAL TRIAL: NCT02169011
Title: Delayed Breast Reconstruction With Skin Flap From the Back
Brief Title: Secondary Breast Reconstruction With a Flap of Skin From the Back
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Collaborators: University of Southern Denmark (Other); Region of Southern Denmark (Other); Sygehus Lillebaelt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-20120207
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Breast Reconstruction
Keywords: Breast reconstruction; Breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Latissimus Dorsi Flap Reconstruction (Active Comparator): Patients are allocated to delayed breast reconstruction with the Latissimus Dorsi flap and if needed an implant.
  Interventions: Procedure: Latissimus Dorsi Flap Reconstruction
- TAP Flap Reconstruction (Active Comparator): Patients are allocated to delayed breast reconstruction with the TAP-flap and if needed an implant in combination with an acellular dermal matrix.
  Interventions: Procedure: TAP Flap Reconstruction

INTERVENTIONS:
Procedure: Latissimus Dorsi Flap Reconstruction — Delayed, unilateral breast reconstruction with the LD-flap. The reconstruction will be performed in a standard fashion as specified in the protocol. Implants should be used when required to gain sufficient volume of the breast.
  Arms: Latissimus Dorsi Flap Reconstruction
Procedure: TAP Flap Reconstruction — Delayed, unilateral breast reconstruction with the TAP-flap. The reconstruction will be performed as specified in the protocol and when implants are required to gain sufficient volume they should be combined with an acellular dermal matrix.
  Arms: TAP Flap Reconstruction

SUMMARY:
The purpose of this study is to examine the different outcomes of breast reconstruction in women who are treated for breast cancer with mastectomy and subsequently have delayed breast reconstruction by one of two different surgical techniques both of which are based on the use of a tissue flap from the patient's back. These techniques are either a latissimus dorsi flap (LD-flap) or a thoracodorsal artery perforator flap (TAP-flap)

The main objective of the study is to establish whether one of these techniques may result in a superior outcome and thus should be recommended as first choice treatment rather than the other.

DETAILED DESCRIPTION:
Women, who are treated for breast cancer with mastectomy, are usually eligible for subsequent reconstruction of the breast. Depending on various conditions the reconstruction can be either immediate or delayed.

Several different surgical techniques for delayed breast reconstruction have been described. An important factor that applies to delayed reconstruction is the lack of excessive, healthy skin in the area where the breast has been removed and the purpose of the surgical techniques developed for this are therefore to provide sufficient amounts of skin and/or other tissues to recreate the contour of the breast. The methods for this can broadly be classified as either expander/implant based or autologous-tissue based. Though full autologous reconstruction is preferred by many surgeons and patients due to the superior result this is not always possible why an implant can be needed in combination with the tissue flap to provide sufficient volume.

In the irradiated patient simple expansion of the skin if often impossible and transfer of autologous tissue is normally required. A wide armamentarium of different methods are available utilizing either pedicled or free flaps for tissue transfer. The most widely used techniques for this in general are reconstruction with abdominal flaps . However, when these women are not eligible for either reconstruction with an abdominal flap or microsurgical reconstruction with other free flaps a well-known and much used technique for reconstruction is the Latissimus Dorsi-flap (LD-flap).

Using this method an island of skin and subcutaneous tissue is provided from the upper part of the patient's back with blood supply deriving from the two main branches of the thoracodorsal artery, which are imbedded in the underlying Latissimus Dorsi muscle. A so called musculocutaneous tissue-flap is raised from the patient's back and tunnelled to the front of the thorax carrying the entire Latissimus Dorsi muscle and the paddle of overlying skin. At the front of the chest the muscle is usually used to drape a silicone implant, and the skin is used to recreate the breast mound. This method is very well-described in the literature, offers a safe and reliable option for breast reconstruction and is often used for this purpose.

Donor site sequelae are however debated. A direct consequence of transferring the Latissimus Dorsi muscle during the procedure is loss of the muscles function in the shoulder and upper arm which involves extension, adduction and rotation of the shoulder joint. Partial impairment in the form of reduced strength and/or restricted movement is thus to be expected as is pain and weakness in the neck, shoulder and upper arm. Other muscles can replace the lost function of the Latissimus Dorsi, and with sufficient rehabilitation and training patients are expected to regain normal function over time. Long term sequelae in the form of chronic pain, discomfort, weakness and/or restricted range of motion have been described but the evidence on this particular area are ambiguous. There are no systematic reviews of the evidence in the published literature and most papers comprise case reports and retrospective cohort studies although a few prospective studies also exist. The different papers indicate varying rates of long-term morbidity associated with the shoulder and arm but the risk of some impairment and chronic pain cannot be ignored based on the available evidence.

At Vejle Hospital in Denmark, we have adopted a new technique for total breast reconstruction as an alternative to the LD-flap in July 2011. This method makes use of a fasciocutaneous flap, which is also raised from the patient's back. Although the blood supply also derives from the Thoracodorsal artery imbedded in the Latissimus Dorsi muscle the flap only contains skin and subcutaneous tissue. The perfusion of blood is instead supplied through a perforator artery, normally arising from the descending branch of the main vessel. This flap is called a Thoracodorsal Artery Perforator-flap (TAP-flap/TDAP-flap) and was first described in the literature in 1995 .

Use of the TAP flap as a pedicled perforator flap have been described in several cases aiding in the treatment of defects on the trunk, upper extremity, head and neck. In the field of breast surgery it has primarily been used for oncoplastic procedures, although a few papers describe the preliminary use of the TAP-flap in combination with an implant for total reconstruction of a breast. As this technique was only recently adopted none of the published studies examine the long term results nor the advantages of using the TAP-flap. A single retrospective study investigates shoulder function after harvest of the flap and finds no affection of the shoulder joint or the upper arm .

We have chosen to perform a modified version of the technique combining the TAP-flap and implant with the use of an acellular dermal matrix (ADM). This matrix is used to drape the lower pole of the implant and in a sense creates an internal bra that supports the prosthesis. We presume that this in part replaces the supportive effect that is normally provided by the muscle when using the LD-flap. The ADM is thus used as a substitute for the patient's own tissue and will over time become integrated as a part of it.

Applying this technique the upper part of the silicone implant is covered by the Major Pectoral muscle, while the lower part is draped by the ADM. The matrix is sutured to the free, lower edge of the muscle as well as to the chest wall at the desired level of the new inframammary fold. This covers and fixates the implant relieving pressure on the flap which is afterwards used to cover the reconstructed mound. We believe this enhances sufficient blood supply to the flap and thus provides the most optimal conditions in terms of obtaining complication-free healing.

Harvest of the TAP-flap allows the Latissimus Dorsi muscle to be left undissected in most cases. When indicated a small cuff of muscle surrounding the dominating perforator can be included in the flap or a small back cut inferiorly to the perforator can be made to allow tension free rotation of the skin paddle. In all cases the procedure is expected to leave the muscle function intact.

Though the TAP flap is well-described for several reconstructive purposes application of the flap as a tool for total breast reconstruction is a new endeavour and its importance has not yet been established. Based on the flaps properties and the more gentle dissection/harvest of the tissue which leaves the underlying Latissimus Dorsi muscle intact we presume the application of this new technique to facilitate a statistically significant reduction in the associated morbidity in terms of impairment and/or chronic pain in the shoulder, back and upper arm which can been experienced after LD-flap based reconstruction.

Furthermore we expect the use of the TAP-flap to cause a decrease in the need for postoperative physical rehabilitation in terms of physiotherapy and training. The aim of this study is thus to test whether this hypothesis is true in order to establish whether the TAP-flap based reconstruction offers any advantages should be favoured above the conventional LD-based reconstruction.

The main objective of this study is to determine whether any detectable difference in shoulder affection distinguishes these two techniques. For this purpose we have designed two separate trials:

Retrospective Follow-up Trial This part of the study intends to examine and compare historical data on women who have already had a delayed breast reconstruction by one of the two methods. The main goal of this pilot study is to collect and analyse all existing information in order to provide a sound background knowledge that should serve as basis for the following RCT. Most importantly this study should provide sufficient data to perform an accurate calculation of the sample size.

Randomized Clinical Trial This trial will be conducted as a confirmatory superiority trial. The intend is to collect, examine and compare data on the two surgical techniques in order to test superiority of the TAP-flap based reconstruction in accordance with our hypothesis as specified above.

The trial is thus designed with two parallel study-arms as patients are allocated to reconstruction by either LD-flap or TAP-flap in the ratio 1:1. As the clinically most important parameter seems to be any objective change in shoulder function this will serve as the primary end-point. Patient reported discomfort/pain as well as the need for physical rehabilitation will also be investigated and analysed as supportive secondary end-points.

In addition to the above data on a number of other patient-related outcomes will be collected as part of this trial. These issues will be addressed as tertiary end-points of a more exploratory nature. We expect these data to supply useful knowledge for further investigations in separate studies.

Designed as multicentre trial patient enrolment and all collection of data will be performed at academic hospitals in Denmark and Norway. All Danish units specializing in plastic and reconstructive surgery who are familiar with both techniques used in this protocol have been invited to participate in this trial. In addition one centre in Skien, Norway, who adopted the TAP-flap technique prior to the initiation of the trial, was invited to participate.

To avoid bias relating to the possible effect on the outcome measures caused by other surgical procedures such as mastectomy and axillary surgery performed simultaneously with the reconstruction only delayed procedures will be studied, as these are also most commonly the cases where autologous tissue transfer is required.

A password protected, electronic database placed on a secure server will be established. This database will only be accessible to the primary investigator and members of the research group who will be involved in the analysis of data. Data are not blinded in relation to allocated treatment.

This study will provide a better knowledge of the expected outcome of delayed breast reconstruction, when it is performed by one of these two surgical techniques. Thus the investigators expect that these results will help determine if the TAP-flap in combination with ADM may represent a better and gentler method for reconstruction of the breast with lower morbidity and better cost-effectiveness than the conventional LD-flap. In all cases the results of this trial will enable us to provide patients with better and more objective information, before they are subjected to delayed breast reconstruction.

ELIGIBILITY:
To avoid bias relating to the possible effect on the outcome measures caused by other surgical procedures such as mastectomy and axillary surgery performed simultaneously with the reconstruction only delayed procedures will be studied, as these are also most commonly the cases where autologous tissue transfer is required.

Patients that should thus be assessed for eligibility will include all women referred to the participating centres for unilateral, delayed breast reconstruction in the inclusion period. The criteria for participation are as follows:

Inclusion criteria:

1) Women over 18 years of age who are referred in the period between 1st of September 2013 and 30st of August 2015 for the purpose of unilateral, delayed breast reconstruction, and who are found best suited for reconstruction with a pedicled tissue flap from the back.

Exclusion criteria

1. Patients found better suited for reconstruction by another method i.e. abdominal or free flap-reconstruction or expander/implant-based reconstruction.
2. Patients with severe dementia that makes it impossible to collect data or obtain informed consent
3. Non-Danish speaking patients from whom informed consent cannot be obtained by interpreter
4. Patients where a suited perforator of the Thoracodorsal artery cannot be identified by colour Doppler ultrasonography.

All women referred for delayed breast reconstruction in the inclusion period will be assessed for eligibility and those meeting the criteria of the study population will be invited to participate in the study. The assessment will be conducted at the preliminary examination in the outpatient clinic by one of the centres consultants assigned to the trial.

Invited patients will receive both oral and written participant information after which a period of minimum 14 days is required before the patient can be enrolled in the trial in accordance with the The Danish Health Act.

Patients considering participation will be invited for a second consultation where written informed consent will be obtained from all who accept the invitation. Randomization will be performed immediately afterwards allocating the patient to reconstruction by either the LD-flap or the TAP-flap. Patients who do not which to be enrolled in the trial will be offered reconstruction with the LD-flap as this must be considered standard of care.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Shoulder Function | 1 year
  The most important difference between the two procedures is the involvement of the muscle and change in shoulder function is the most relevant clinical measure to investigate.
  For evaluation of shoulder function we use the internationally validated Constant Shoulder Score (CSS). This system assess pain, function in everyday-life, range of motion and strength and incorporates these parameters into one total score. It is the recommended scoring-system by the European Society of Shoulder and Elbow Surgery. Each variable in the system is evaluated separately.
  For all patients scoring will be performed preoperatively as well as 3, 6 and 12 months postoperatively. Shoulder function will be evaluated bilaterally at all stages. To avoid multiplicity-issues the primary end-point has been defined as the difference in the total score between the baseline evaluation preoperatively and the evaluation one year postoperatively.

SECONDARY OUTCOMES:
Patient Reported Discomfort | 1 year
  As the pain-related outcome measure in the CSS only concerns pain in the shoulder an assessment of the patients experience of pain and/or tightening in the neck, back, arm or breast will be performed at baseline and 3, 6 and 12 months postoperatively. For this the following frasing will be used:
  "Have you experienced either pain, tightening or discomfort in your neck, back, arm or the reconstructed breast during the last month?"
  All patients indicating any symptomatology will be asked the following:
  "On a scale from 1-10, where 1 indicates the lowest level of pain or discomfort and 10 the highest, please indicate the worst level of pain or discomfort you have experienced in the past month"
  A median value of the level of discomfort at each time-point will be calculated for each patient-group and tested for statistically significant difference as the most important supportive secondary end-points.
Rehabilitation | 1 year
  The patients need for physical rehabilitation and training will be addressed as the second most important supportive secondary end-point.
  A patient reported quantification of the time spent weekly on either physiotherapy or training targeted on the shoulder, arm and/or back will be made at baseline. All patients will follow the same rehabilitation program in the postoperative phase and for the first 3 months after surgery. Hereafter the rehabilitation will be individual and based on their specific needs.
  As for evaluation of the shoulder function, registration of average time spent weekly on physiotherapy/training will be made by the primary investigator in the outpatient clinic 6 and 12 months postoperatively. A median value of the time spent weekly on physiotherapy and shoulder-specific training at each time-point will be calculated for each patient-group and tested for statistically significant difference as supportive secondary end-points.

OTHER OUTCOMES:
Quality-of-life | 1 year
  The patients' quality-of-life will be assessed before and after reconstruction using the international validated questionnaire developed The European Organisation for Research and Treatment of Cancer (EORTC) for assessment of life quality in cancer patients. Patients will be asked to complete the general questionnaire QLQ-30 in combination with the additional questionnaire QLQ-BR23 that has been specifically developed for cancer patients with breast-related diseases . The questionnaires will be completed in the outpatient clinic preoperatively and again 12 months after surgery.
Socio-economics | 1 year
  In order to evaluate the socio-economic aspects and cost-benefit associated with the use of each surgical technique we record the following parameters for all patients: Duration of operation, duration of hospitalization, duration of entire course of the breast reconstruction, duration of sick leave and need for revisional/correctional procedures. Based on the data collected we will perform an evaluation of the total expenditure associated with the two different types of delayed reconstruction. This evaluation will comprise an estimate of the costs associated with the procedures including expenses for utensils, implants and ADM as well as an estimate of the expenses related to hospitalization, sick leave and rehabilitation.
Aesthetic Outcome | 1 year
  We wish to conduct an evaluation of the aesthetic result of the different reconstructions including a professional assessment and an assessment from the patient. Hence all patients will be asked to evaluate the appearance of their bosom on a scale from 1 to 10 indicating their satisfaction with the reconstruction.
  Furthermore the patients will be subjected to a professional evaluation as all women will have their bosom photographed. Photographs will be evaluated by two unbiased medical consultants specializing in plastic surgery who are not associated with the department or the project. These specialists will be asked to perform the same evaluation as the patients.
  Both the patient's and the specialist's evaluation will be performed before surgery and once again at the final consultation in the outpatient clinic 12 months following the reconstruction.
Complications | 3 months
  Complications following the surgery will be recorded continuously during hospitalization and in the outpatient's clinic. They will include: skin necrosis and/or delayed healing, infection, seromas, bleeding, flap-necrosis and explantation. Complications will be classified as either major or minor depending on the need for surgical revision.

CONTACTS AND LOCATIONS:
Overall Officials: Jørn B Thomsen, MD, PhD, Study Chair — Center Hospital Lillebaelt, Institute of Regional Health Research, University of Southern Denmark
Locations (4):
- Denmark (3):
  - Herlev Hospital, Herlev
  - Odense University Hospital, Odense
  - Vejle Hospital, Vejle
- Telemark Hospital, Skien, Telemark, Norway

REFERENCES:
- [Background] Bonomi S, Settembrini F, Salval A, Gregorelli C, Musumarra G, Rapisarda V. Current indications for and comparative analysis of three different types of latissimus dorsi flaps. Aesthet Surg J. 2012 Mar;32(3):294-302. doi: 10.1177/1090820X12437783. PMID 22395320
- [Background] Perdikis G, Koonce S, Collis G, Eck D. Latissimus dorsi myocutaneous flap for breast reconstruction: bad rap or good flap? Eplasty. 2011;11:e39. Epub 2011 Oct 17. PMID 22031843
- [Background] Garusi C, Lohsiriwat V, Brenelli F, Galimberti VE, De Lorenzi F, Rietjens M, Rossetto F, Petit JY. The value of latissimus dorsi flap with implant reconstruction for total mastectomy after conservative breast cancer surgery recurrence. Breast. 2011 Apr;20(2):141-4. doi: 10.1016/j.breast.2010.10.007. Epub 2010 Nov 11. PMID 21074437
- [Background] Hammond DC. Latissimus dorsi flap breast reconstruction. Plast Reconstr Surg. 2009 Oct;124(4):1055-1063. doi: 10.1097/PRS.0b013e3181b6bf05. PMID 19935289
- [Background] Dejode M, Bordes V, Jaffre I, Classe JM, Dravet F. [Oncologic, functional, and aesthetics results; evaluation of the quality of life after latissimus dorsi flap breast reconstruction. About a retrospective series of 450 patients]. Ann Chir Plast Esthet. 2011 Jun;56(3):207-15. doi: 10.1016/j.anplas.2011.01.003. Epub 2011 Mar 29. French. PMID 21450385
- [Background] Forthomme B, Heymans O, Jacquemin D, Klinkenberg S, Hoffmann S, Grandjean FX, Crielaard JM, Croisier JL. Shoulder function after latissimus dorsi transfer in breast reconstruction. Clin Physiol Funct Imaging. 2010 Nov;30(6):406-12. doi: 10.1111/j.1475-097X.2010.00956.x. PMID 20633032
- [Background] Faucher A, Barrault M, Duguey I. [Contribution to the study of painful and functional sequellae after breast reconstruction using latissimus dorsi flap. Investigation into 149 patients]. Ann Chir Plast Esthet. 2010 Apr;55(2):104-10. doi: 10.1016/j.anplas.2009.04.008. Epub 2009 Oct 29. French. PMID 19879032
- [Background] Button J, Scott J, Taghizadeh R, Weiler-Mithoff E, Hart AM. Shoulder function following autologous latissimus dorsi breast reconstruction. A prospective three year observational study comparing quilting and non-quilting donor site techniques. J Plast Reconstr Aesthet Surg. 2010 Sep;63(9):1505-12. doi: 10.1016/j.bjps.2009.08.017. Epub 2009 Oct 12. PMID 19819774
- [Background] Koh CE, Morrison WA. Functional impairment after latissimus dorsi flap. ANZ J Surg. 2009 Jan-Feb;79(1-2):42-7. doi: 10.1111/j.1445-2197.2008.04797.x. PMID 19183378
- [Background] Glassey N, Perks GB, McCulley SJ. A prospective assessment of shoulder morbidity and recovery time scales following latissimus dorsi breast reconstruction. Plast Reconstr Surg. 2008 Nov;122(5):1334-1340. doi: 10.1097/PRS.0b013e3181881ffe. PMID 18971716
- [Background] Adams WP Jr, Lipschitz AH, Ansari M, Kenkel JM, Rohrich RJ. Functional donor site morbidity following latissimus dorsi muscle flap transfer. Ann Plast Surg. 2004 Jul;53(1):6-11. doi: 10.1097/01.sap.0000106430.56501.b5. PMID 15211190
- [Background] Hamdi M, Van Landuyt K, Hijjawi JB, Roche N, Blondeel P, Monstrey S. Surgical technique in pedicled thoracodorsal artery perforator flaps: a clinical experience with 99 patients. Plast Reconstr Surg. 2008 May;121(5):1632-1641. doi: 10.1097/PRS.0b013e31816c3bfa. PMID 18453987
- [Background] Hamdi M, Salgarello M, Barone-Adesi L, Van Landuyt K. Use of the thoracodorsal artery perforator (TDAP) flap with implant in breast reconstruction. Ann Plast Surg. 2008 Aug;61(2):143-6. doi: 10.1097/SAP.0b013e318158fd7b. PMID 18650605
- [Background] Hamdi M, Decorte T, Demuynck M, Defrene B, Fredrickx A, Maele GV, De Pypere H, Landuyt KV, Blondeel P, Vanderstraeten G, Monstrey S. Shoulder function after harvesting a thoracodorsal artery perforator flap. Plast Reconstr Surg. 2008 Oct;122(4):1111-1117. doi: 10.1097/PRS.0b013e31818459b4. PMID 18827644
- [Background] Sbitany H, Serletti JM. Acellular dermis-assisted prosthetic breast reconstruction: a systematic and critical review of efficacy and associated morbidity. Plast Reconstr Surg. 2011 Dec;128(6):1162-1169. doi: 10.1097/PRS.0b013e318230c29e. PMID 22094735
- [Background] Hoppe IC, Yueh JH, Wei CH, Ahuja NK, Patel PP, Datiashvili RO. Complications following expander/implant breast reconstruction utilizing acellular dermal matrix: a systematic review and meta-analysis. Eplasty. 2011;11:e40. Epub 2011 Nov 3. PMID 22084645
- [Background] Himsl I, Drinovac V, Lenhard M, Stockl D, Weissenbacher T, Dian D. The use of porcine acellular dermal matrix in silicone implant-based breast reconstruction. Arch Gynecol Obstet. 2012 Jul;286(1):187-92. doi: 10.1007/s00404-012-2266-x. Epub 2012 Mar 2. PMID 22382372
- [Background] Heneghan HM, Prichard RS, Lyons R, Regan PJ, Kelly JL, Malone C, McLaughlin R, Sweeney KJ, Kerin MJ. Quality of life after immediate breast reconstruction and skin-sparing mastectomy - a comparison with patients undergoing breast conserving surgery. Eur J Surg Oncol. 2011 Nov;37(11):937-43. doi: 10.1016/j.ejso.2011.08.126. Epub 2011 Sep 6. PMID 21899982
- [Background] Metcalfe KA, Semple J, Quan ML, Vadaparampil ST, Holloway C, Brown M, Bower B, Sun P, Narod SA. Changes in psychosocial functioning 1 year after mastectomy alone, delayed breast reconstruction, or immediate breast reconstruction. Ann Surg Oncol. 2012 Jan;19(1):233-41. doi: 10.1245/s10434-011-1828-7. Epub 2011 Jun 15. PMID 21674270
- [Background] Bellino S, Fenocchio M, Zizza M, Rocca G, Bogetti P, Bogetto F. Quality of life of patients who undergo breast reconstruction after mastectomy: effects of personality characteristics. Plast Reconstr Surg. 2011 Jan;127(1):10-17. doi: 10.1097/PRS.0b013e3181f956c0. PMID 21200194
- [Background] Freitas-Silva R, Conde DM, de Freitas-Junior R, Martinez EZ. Comparison of quality of life, satisfaction with surgery and shoulder-arm morbidity in breast cancer survivors submitted to breast-conserving therapy or mastectomy followed by immediate breast reconstruction. Clinics (Sao Paulo). 2010 Jun;65(8):781-7. doi: 10.1590/s1807-59322010000800007. PMID 20835555
- [Background] Gahm J, Wickman M, Brandberg Y. Bilateral prophylactic mastectomy in women with inherited risk of breast cancer--prevalence of pain and discomfort, impact on sexuality, quality of life and feelings of regret two years after surgery. Breast. 2010 Dec;19(6):462-9. doi: 10.1016/j.breast.2010.05.003. Epub 2010 Jun 3. PMID 20605453
- [Background] Wasteson E, Sandelin K, Brandberg Y, Wickman M, Arver B. High satisfaction rate ten years after bilateral prophylactic mastectomy - a longitudinal study. Eur J Cancer Care (Engl). 2011 Jul;20(4):508-13. doi: 10.1111/j.1365-2354.2010.01204.x. Epub 2010 Jun 29. PMID 20597955
- [Background] Min SY, Kim HY, Jung SY, Kwon Y, Shin KH, Lee S, Kim SW, Kang HS, Yun YH, Lee ES. Oncological safety and quality of life associated with mastectomy and immediate breast reconstruction with a latissimus dorsi myocutaneous flap. Breast J. 2010 Jul-Aug;16(4):356-61. doi: 10.1111/j.1524-4741.2010.00941.x. Epub 2010 Jun 10. PMID 20545939
- [Background] Atisha D, Alderman AK, Lowery JC, Kuhn LE, Davis J, Wilkins EG. Prospective analysis of long-term psychosocial outcomes in breast reconstruction: two-year postoperative results from the Michigan Breast Reconstruction Outcomes Study. Ann Surg. 2008 Jun;247(6):1019-28. doi: 10.1097/SLA.0b013e3181728a5c. PMID 18520230
- [Background] Constant CR, Gerber C, Emery RJ, Sojbjerg JO, Gohlke F, Boileau P. A review of the Constant score: modifications and guidelines for its use. J Shoulder Elbow Surg. 2008 Mar-Apr;17(2):355-61. doi: 10.1016/j.jse.2007.06.022. Epub 2008 Jan 22. No abstract available. PMID 18218327
- [Background] Pacella SJ, Vogel JE, Locke MB, Codner MA. Aesthetic and technical refinements in latissimus dorsi implant breast reconstruction: a 15-year experience. Aesthet Surg J. 2011 Feb;31(2):190-9. doi: 10.1177/1090820X10395506. PMID 21317117
- [Background] Wirth R, Banic A, Erni D. Aesthetic outcome and oncological safety of nipple-areola complex replantation after mastectomy and immediate breast reconstruction. J Plast Reconstr Aesthet Surg. 2010 Sep;63(9):1490-4. doi: 10.1016/j.bjps.2009.08.014. Epub 2009 Oct 4. PMID 19805012
- [Background] Gahm J, Jurell G, Edsander-Nord A, Wickman M. Patient satisfaction with aesthetic outcome after bilateral prophylactic mastectomy and immediate reconstruction with implants. J Plast Reconstr Aesthet Surg. 2010 Feb;63(2):332-8. doi: 10.1016/j.bjps.2008.11.014. Epub 2008 Dec 13. PMID 19071075
- [Derived] Makki A, Thomsen JB, Gunnarsson GL, Holmich PLR, Sorensen PJA, Rindom MB. A cost-effectiveness analysis of delayed breast reconstruction with pedicled flaps from the back. J Plast Reconstr Aesthet Surg. 2022 Jul;75(7):2211-2218. doi: 10.1016/j.bjps.2022.02.034. Epub 2022 Feb 26. PMID 35365412